CLINICAL TRIAL: NCT04638465
Title: De-Escalation Protocol Of HPV Mediated Oropharyngeal Squamous Cell Carcinoma Based On The AJCC 8th Edition Staging Manual
Brief Title: De-Escalation Protocol Of HPV Mediated Oropharyngeal Squamous Cell Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Nebraska Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: MECC-HN01
Record Dates: First submitted 2020-11-11; First posted 2020-11-20 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-04

CONDITIONS: HPV-Mediated (P16-Positive) Oropharyngeal Carcinoma by AJCC V8 Clinical Stage; Oropharynx Cancer
Keywords: HPV-Mediated; Oropharyngeal Cancer; P16-Positive
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- A - Surgery Only: Participants with the following diagnosis will receive transoral robotic surgery with neck dissection:
  * Base of Tongue/Non-Tonsil Oropharynx - Stage: cT1-2, cN0 or N1 (single node)
  * Tonsil - Stage: cT1-3, cN0 or N1 (single node)
  * Unknown primary - Stage: cT0 N1 (single node)
  Radiation also given if indicated by intermediate or high risk features following surgery.
  Interventions: Procedure: Transoral robotic surgery
- B - Surgery with Adjuvant Therapy: Participants with the following diagnosis will receive surgery followed by 6 Cycles of Cisplatin 40 mg/m2:
  * Base of Tongue/Non-Tonsil Oropharynx - Stage: cT1-2, cN1 (2-4 nodes) or N2
  * Tonsil - Stage: cT1-3, N1 (2-4 nodes)
  Radiation also given if indicated by intermediate or high risk features following surgery.
  Interventions: Procedure: Transoral robotic surgery; Drug: Cisplatin - Dose Level 1
- C - Concurrent Chemo/Radiation Therapy - Dose Level 1: Participants with the following diagnosis will receive 6 Cycles of Cisplatin 40 mg/m2 + 60 Gy Radiation:
  * Tonsil - Stage: cT1-3, N2
  * Unknown Primary - Stage: cT0, N2
  Interventions: Drug: Cisplatin - Dose Level 1; Radiation: Dose Level 1
- D - Concurrent Chemo/Radiation Therapy - Dose Level 2: Participants with the following diagnosis will receive 7 Cycles of Cisplatin 40 mg/m2 + 70 Gy Radiation:
  * Base of Tongue/Non-Tonsil Oropharynx - Stage: cT3-4, any N
  * Base of Tongue/Non-Tonsil Oropharynx - Stage: cAny T, N3
  * Tonsil - Stage: cT1-3, N3
  * Tonsil - Stage: cT4, any N
  * Unknown Primary - Stage: cT0, N3
  Interventions: Drug: Cisplatin - Dose Level 2; Radiation: Dose Level 2

INTERVENTIONS:
Procedure: Transoral robotic surgery — Transoral resection with neck dissection
  Groups: A - Surgery Only; B - Surgery with Adjuvant Therapy
Drug: Cisplatin - Dose Level 1 — 6 Cycles of 40 mg/m2
  Groups: B - Surgery with Adjuvant Therapy; C - Concurrent Chemo/Radiation Therapy - Dose Level 1
Drug: Cisplatin - Dose Level 2 — 7 Cycles of 40 mg/m2
  Groups: D - Concurrent Chemo/Radiation Therapy - Dose Level 2
Radiation: Dose Level 1 — 60 Gy/6 weeks - 2 Gy/fraction, 5 fractions/week
  Groups: C - Concurrent Chemo/Radiation Therapy - Dose Level 1
Radiation: Dose Level 2 — 70 Gy/7 weeks - 2 Gy/fraction, 5 fractions/week
  Groups: D - Concurrent Chemo/Radiation Therapy - Dose Level 2

SUMMARY:
The purpose of this study is to evaluate the effects, good and/or bad, of treating participants with HPV-mediated oropharyngeal cancer, with less treatment, using the new staging system. The investigators believe this treatment will provide the same effectiveness as the usual treatment, but decrease the side effects. The radiation doses, chemotherapy doses, and the type of surgical approaches that will be used in this treatment protocol have all been previously investigated. Previous research suggests that this can be done safely, but there has not been a study done basing treatment on the new staging system.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have newly diagnosed, histologically, or cytologically confirmed HPV positive, squamous cell carcinoma of the base of tongue, tonsil, oropharyngeal cavity or unknown primary.
* Participants must have tumors staged using AJCC TNM 8th edition Staging for Head and Neck cancers.
* Participants must have an exam by a Head and Neck Oncologist within 6 weeks before registration.
* Participants must not have any evidence of distant metastatic disease.
* Participants with other active malignancies may be eligible, at the discretion of the investigator, as long as the treatment plan for the head and neck cancer outlined in this protocol can still be followed. The potential effect of the treatment and disease progress of the second active malignancy should also have minimal or no impact on the toxicities being monitored on this study.
* Participants must not have any uncontrolled intercurrent illnesses, psychiatric illnesses, psychosocial problems, or social situations that would limit the patient's compliance with the study or ability to successfully complete the study treatment safely.
* Participants with inconclusive pathology after biopsy; who are found to have HPV positive SCC following standard of care surgery are eligible to enroll.
* Participants who require additional surgery to complete staging with known HPV+ SCC are eligible to enroll.

Exclusion Criteria:

* Participants must not be receiving or planning to receive any other clinical trial therapy or intervention.
* Participants with an unknown primary tumor who are both HPV positive and EBV positive are NOT eligible for this protocol.

These additional evaluations must be performed on participants with T0 (unknown primary site) P16+ squamous cell carcinoma of the head and neck prior to registration.

* Flexible laryngoscope
* Ultrasound guided Fine-needle aspirate (FNA) of the known site of disease with the following analysis:
* Human papilloma virus (HPV); p16 Immuno-Histo-Chemical Staining. If negative, complete high risk HPV Fluorescence in-situ Hybridization (FISH).
* Epstein Barr Virus (EBV): Epstein Barr Virus Encoded RNA (EBER) in-situ Hybridization.
* Direct Laryngoscopy with directed biopsy of bilateral base of tongue, bilateral palatine tonsillectomy, and dental extraction, as needed.

If a participant is both HPV positive and EBV positive, he/she is not eligible.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have newly diagnosed, histologically, or cytologically confirmed HPV positive, squamous cell carcinoma of the base of tongue, tonsil, oropharyngeal cavity or unknown primary. Participants must have tumors staged using AJCC TNM 8th edition Staging for Head and Neck cancers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From randomization to death, assessed up to 10 years
  To determine if overall survival remains the same with the de-escalated protocol as the historical standard of care survival benefit.
Disease Free Survival | From randomization to date of progression, second primary tumor from the head and neck region, or death, assessed up to 10 years
  To determine if disease free survival remains the same with the de-escalated protocol as the historical standard of care survival benefit.

SECONDARY OUTCOMES:
Rate of Patients with a Grade 3 or Higher Adverse Event | From randomization to death, assessed up to 10 years
  To evaluate the side effects patients experience when being treated on the de-escalated protocol.
Measure the quality of life of participants using the FACT H&N assessment tool | From randomization to death, assessed up to 10 years
  To evaluate the quality of life of patients who are treated with the de-escalated protocol.
Measure the depression of participants using the Self-Report Quick Inventory of Depressive Symptomatology assessment | From randomization to death, assessed up to 10 years
  To evaluate depression in patients who are treated with the de-escalated protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Nebraska Methodist Hospital, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Panwar A, Shah S, Reid AE, Lydiatt W, Holcomb AJ, Osmolak A, Coughlin A, Militsakh O, Su YB, Mirmiran A, Huang TS, Nolan N, Duckert R, Barney C, Chiu M, Nguyen C, Sayles H, Ganti AK, Lindau R. Quality of Life and Depression Symptoms After Therapy De-Escalation in HPV+ Oropharyngeal Squamous Cell Carcinoma: A Nonrandomized Controlled Trial. JAMA Otolaryngol Head Neck Surg. 2024 May 1;150(5):429-435. doi: 10.1001/jamaoto.2024.0262. PMID 38573597